CLINICAL TRIAL: NCT00759083
Title: Bivalirudin PCI Registry in HIT/HITTS Patients
Brief Title: Bivalirudin PCI Registry in Heparin Induced Thrombocytopenia/Heparin Induced Thrombocytopenia and Thrombosis Syndrome (HIT/HITTS) Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was discontinued early due to inadequate patient enrollment. No patients were enrolled.
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TMC-BIV-07-02
Record Dates: First submitted 2008-09-22; First posted 2008-09-25 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Heparin-Induced Thrombocytopenia; Heparin-induced Thrombocytopenia and Thrombosis Syndrome
Keywords: HIT; HITTS
MeSH Terms: interventions — bivalirudin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Patients with HIT/HITTS who require anticoagulation for PCI
  Interventions: Drug: bivalirudin

INTERVENTIONS:
Drug: bivalirudin — Bivalirudin; 0.75mg/kg/h IV bolus followed immediately by 1.75 mg/kg/h infusion for the duration of the procedure

SUMMARY:
To monitor the frequency of the development of thrombocytopenia in patients with Heparin Induced Thrombocytopenia/Heparin Induced Thrombocytopenia and Thrombosis Syndrome receiving bivalirudin during Percutaneous Coronary Intervention

ELIGIBILITY:
Inclusion Criteria:

* Clinically Documented History of HIT/HITTS
* Suspicion of HIT/HITTS

Exclusion Criteria:

* Bleeding Diathesis
* Ischemic Stroke
* Chronic Thrombocytopenia
* Hematologic Malignancy
* Contraindication to bivalirudin
* Pregnant or nursing mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual); Study Completion 2010-05-10 (Actual)

PRIMARY OUTCOMES:
Platelet counts | 6, 12, 24, 48 Hours

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Ohman, MD, Principal Investigator — Duke Clinical Research Institute
Locations (1):
- Duke Clinical Research Institute, Durham, North Carolina, United States